CLINICAL TRIAL: NCT02125149
Title: Prenatal Physical Activity Intervention
Brief Title: The Expecting Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202954
Record Dates: First submitted 2014-04-21; First posted 2014-04-29 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy; Obese
Keywords: pregnancy; obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard of care
- Intervention (Experimental): Exercise intervention from 12 week gestation until delivery
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention
  Arms: Intervention

SUMMARY:
The purpose of the study is to determine how a mother's health and physical activity may influence her child's growth and development.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30
* >18 years of age
* Singleton pregnancy
* Less than 12 weeks gestation
* Sedentary
* Conceived without assisted fertility treatments
* Cleared by physician to exercise

Exclusion Criteria:

* Women with pre-existing medical conditions as determined by the PI to affect the outcomes of interest
* Women who are using recreational drugs, tobacco, or alcohol during pregnancy
* Women with contraindications to exercise during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2014-09-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Risk of obesity in infants and children | 2 years
  Birth weight, body fat, and metabolism will be evaluated during the first 2 years of life.

SECONDARY OUTCOMES:
Maternal insulin sensitivity | 9 months
  Fasted blood samples will be analyzed to assess glucose and insulin.
Maternal inflammation | 9 months
  Markers of inflammation will be investigated in fasted serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, Ph.D, Principal Investigator — UAMS
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Saben JL, Sims CR, Piccolo BD, Andres A. Maternal adiposity alters the human milk metabolome: associations between nonglucose monosaccharides and infant adiposity. Am J Clin Nutr. 2020 Nov 11;112(5):1228-1239. doi: 10.1093/ajcn/nqaa216. PMID 32844207